CLINICAL TRIAL: NCT02308657
Title: A Multicenter Observational Study to Assess the Variability of Molecular Biomarkers and Clinical Measures in Patients With Myotonic Dystrophy Type 1
Brief Title: Multicenter Observational Study of Myotonic Dystrophy Type 1
Acronym: MOS-DM1/POP
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: University of Florida (Other); University of Kansas Medical Center (Other); Ohio State University (Other); Stanford University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Biogen (Industry); Muscular Dystrophy Association (Other); Myotonic Dystrophy Foundation (Other); The Marigold Foundation (Unknown)
Responsible Party: Principal Investigator, Charles Thornton, Principal Investigator, University of Rochester
Other Study IDs: RSRB48991; U54NS048843 (NIH); NCT02176798 (obsolete NCT alias)
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-02

CONDITIONS: Myotonic Dystrophy Type 1
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be used for routine laboratory testing, such as tests of blood cells, chemistry, and ability to form blood clots. Blood samples will be used for genetic testing (DNA testing) and to identify biomarkers. Needle muscle biopsies will be obtained from the tibialis anterior, a muscle in the front of the leg, next to the shin.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to determine the best ways to assess how people are affected by myotonic dystrophy type 1 (DM1). The study will assess walking speed, muscle strength, muscle size, myotonia, heart rhythm, mental efficiency, and overall health. Participants will complete questionnaires to record their ideas about how they are affected by DM1. The study will evaluate people with DM1 over 1 year to determine how the condition changes over time. The study will identify biomarkers of DM1. Biomarkers are laboratory measurements that show the effects of DM1 on a person's muscle tissue or blood. Biomarkers are needed in future studies to determine how DM1 may respond to treatments.

DETAILED DESCRIPTION:
Participants in the study will come to the study site for 3 study visits. Each visit will take most of the day. Each visit will include a series of evaluations to determine how the person is affected by myotonic dystrophy. The results from the initial study visit will be compared to the second study visit after 3 months and the third study visit after 1 year. A small needle biopsy of a leg muscle will be performed at the first and second study visits (but not at the third visit). After the second study visit, participants will be asked to make a phone call every day for 30 days to report their symptoms and muscle strength (grip strength).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed informed consent and authorization to use protected health information in accordance with national and local patient privacy regulations.
* Men and women, 18 to 70 years old, inclusive; body mass index ≤33.
* Onset of DM1 after age 10.
* Clinical diagnosis of DM1 based on research criteria or prior genetic testing with confirmation of CTG repeat length ≥70. A genetic test confirming DM1 is not required for entry. A DNA sample will be obtained from all subjects for DM1 genetic testing. If this test does not show an expanded repeat in the DM1 gene the subject will be withdrawn from the study.
* Ability to complete a 6 minute walk test (ankle-foot braces are allowed, but cane and walker are not allowed).

Exclusion Criteria:

* Clinically significant infections or medical illness from 30 days prior to Visit 1.
* History of, or abnormal laboratory values indicative of, significant medical, neurologic (other than DM1), or psychiatric disorders that might preclude participation in the study in the opinion of the Investigator.
* A recent history of any of the following conditions on routine blood screening: white blood cells <3000, platelets <100,000, hematocrit <30%, symptomatic liver disease with serum albumin <3 g/L, or creatinine >1.5 mg%.
* Any of the following medical conditions: uncontrolled or insulin dependent diabetes mellitus, congestive heart failure, symptomatic cardiomyopathy, symptomatic coronary artery disease, cancer (other than skin cancer) within the prior 5 years, multiple sclerosis, or other serious medical illness.
* Myotonic dystrophy type 2 or other diseases that mimic the signs or symptoms of DM1. Coexistence of other neuromuscular disease.
* Thyroid dysfunction that is untreated (if on thyroid hormone replacement therapy, need to have adequate and stable replacement over the previous 6 months).
* Second or third degree heart block, atrial flutter, atrial fibrillation, ventricular tachycardia, or is receiving medication for the treatment of cardiac arrhythmia.
* Liver or kidney disease requiring ongoing treatment.
* Have a seizure disorder.
* Drug or alcohol abuse within 3 months of Visit 1.
* Women who are pregnant or who plan to become pregnant during the study's duration.
* Treatment with supplemental anabolic hormones (including testosterone, human recombinant growth hormone, human recombinant insulin like growth factor-1, other anabolic drug mixtures) during the previous 12 months.
* History of bleeding tendency or ongoing oral anticoagulation.
* Hypersensitivity to local anesthetics or components thereof to be used in the biopsy procedure.
* Participation in any investigational treatment study within 6 months prior to Visit 1.
* Inability or unwillingness to undergo any of the study-specific procedures or assessments, including needle muscle biopsies.
* Medical or other unspecified reasons that in the opinion of the Investigator makes the patient unsuitable for enrollment.
* Treatment with any of the following anti-myotonia medications within 8 weeks prior to Visit 1: phenytoin, carbamazepine, procainamide, disopyramide, nifedipine, acetazolamide, clomipramine, imipramine, mexiletine
* Treatment with corticosteroids within 8 weeks prior to Visit 1.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 100 adult patients (18 to 70 years old, inclusive) with DM1 will be enrolled at 6 centers.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-11; Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Needle Muscle Biopsy RNA Biomarkers | Baseline, 3 months
  To evaluate the stability of RNA splice events as biomarkers of DM1.

SECONDARY OUTCOMES:
Myotonia | Baseline, 3 months, 1 year
  Muscle relaxation time of the hand grip and electromyography (EMG) of a leg muscle (tibialis anterior)
Muscle Strength | Baseline, 3 months, 1 year
  Computer-assisted and manual testing of muscle strength
Myotonic Dystrophy Health Index (MDHI) | Baseline, 3 months, 1 year
  Patient perceptions of their disease burden as measured by a questionnaire.

OTHER OUTCOMES:
Timed functional tests | Baseline, 3 months, 1 year
  Timed functional tests include walking speed, rising from a chair, and climbing steps

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Thornton, MD, Principal Investigator — University of Rochester
Locations (6):
- United States (6):
  - Stanford University, Stanford, California
  - University of Florida, Gainesville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - NIH, Bethesda, Maryland
  - University of Rochester, Rochester, New York
  - Ohio State University, Columbus, Ohio